CLINICAL TRIAL: NCT04532788
Title: Efficacy of Customized Corneal Cross-linking Versus Standard Corneal Cross-linking in Patients With Progressive Keratoconus
Brief Title: Efficacy of Customized Corneal Cross-linking vs. Standard Corneal Cross-linking
Acronym: C-CROSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL73003.068.20
Record Dates: First submitted 2020-08-20; First posted 2020-08-31 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2023-03

CONDITIONS: Keratoconus
Keywords: Keratoconus; Crosslinking; Customized
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Customized crosslinking (Active Comparator): In the customized corneal cross-linking protocol (cCXL) a patient-specific treatment pattern, based on the patient's Pentacam images, will be used to treat the cornea. The CXL pattern exists out of 3 concentric circles and is centered on the cone. To estimate the cone location a combination of the thinnest corneal point, maximum anterior elevation and maximum posterior elevation is used. The epithelium is debrided with alcohol within the marked zone. After the application of riboflavin each circle receives a different amount of energy, which gradually decreases with increasing circle size.
  The procedure is done with the Avedro Mosaic CXL device (Avedro, Inc. Waltham, Massachusetts, United States).
  Interventions: Procedure: Customized crosslinking
- Standard crosslinking (Active Comparator): In the standard corneal cross-linking protocol (sCXL) the epithelium is debrided with alcohol over a region with a diameter of 9.0 mm. After the application of riboflavin the cornea is irradiated with UVA with a fluence of 10 mW/cm2 during 9 minutes with a diameter of 9.0 mm, resulting in a total energy of 5.4 J/cm2.
  The procedure is done with the Avedro Mosaic CXL device (Avedro, Inc. Waltham, Massachusetts, United States).
  Interventions: Procedure: Standard crosslinking

INTERVENTIONS:
Procedure: Customized crosslinking — In the customized corneal cross-linking protocol (cCXL) a patient-specific treatment pattern, based on the patient's Pentacam images, will be used to treat the cornea. The CXL pattern exists out of 3 concentric circles and is centered on the cone. To estimate the cone location a combination of the thinnest corneal point, maximum anterior elevation and maximum posterior elevation is used. The epithelium is debrided with alcohol within the marked zone. After the application of riboflavin each circle receives a different amount of energy, which gradually decreases with increasing circle size.
  The procedure is done with the Avedro Mosaic CXL device (Avedro, Inc. Waltham, Massachusetts, United States).
  Arms: Customized crosslinking
Procedure: Standard crosslinking — In the standard corneal cross-linking protocol (sCXL) the epithelium is debrided with alcohol over a region with a diameter of 9.0 mm. After the application of riboflavin the cornea is irradiated with UVA with a fluence of 10 mW/cm2 during 9 minutes with a diameter of 9.0 mm, resulting in a total energy of 5.4 J/cm2.
  The procedure is done with the Avedro Mosaic CXL device (Avedro, Inc. Waltham, Massachusetts, United States).
  Arms: Standard crosslinking

SUMMARY:
The standard or Dresden protocol was established in 2003 and treats the entire cornea. However, recent ultra-structural research showed that keratoconus is localized. Therefore, treating only the affected zone and minimalizing the risk of damaging surrounding tissues would be beneficial.

The objective of this study is to evaluate whether the effectiveness of customized cross-linking (cCXL) is non-inferior to standard accelerated cross-linking (sCXL) in terms of flattening of the cornea and halting keratoconus progression.

DETAILED DESCRIPTION:
In 2003 Wollensak et al used corneal cross-linking (CXL) in humans to halt the progression of keratoconus. During the procedure the top layer of the cornea, the epithelium, is debrided. Then the cornea is soaked with riboflavin, a photosensitizer. Hereafter a 9.0 mm diameter Ultraviolet-A (UVA) beam radiates the cornea for 30 minutes with a fluence of 3 mW/cm2 resulting in a total energy of 5,4 J/cm2. This protocol is called the Dresden protocol. Currently, accelerated versions of the Dresden protocol are used in common practice. There are different accelerated protocols with fluences of 9mW/cm2, 10mW/cm2 and 15 mW/cm2. The higher the fluence, the shorter the treatment time, however according to the Bunsen-Roscoe reciprocity law the total amount of energy stays the same.During the procedure oxygen radicals are formed that interact with the surrounding molecules, leading to the formation of new chemical bounds between the collagen fibrils (i.e. corneal crosslinks). The final goal of the procedure is to cause the cornea to stiffen and achieve flattening of the treated region.

For any treatment, it is imperative that the unaffected region of the tissue is not unnecessarily treated by an intervention or drug application. To minimalize the risk of damage to surrounding tissues it would be beneficial that the UVA beam is restricted to the affected, keratoconic zone in the patient's cornea. This can be achieved by customizing the beam shape and size in a way that only the degenerated zone is treated, i.e. by customized cross-linking (cCXL). Recently published studies provide clinical evidence that similar clinical outcomes (amount of corneal flattening) can be achieved when only the cone is treated instead of the entire cornea.They also show the potential benefits of cCXL, e.g. the treatment is patient-specific, a smaller surface of the cornea is irradiated, lower incidence of corneal haze, a faster reepithelialisation and a shorter procedure time. However, none of these studies are randomized and study results are limited by using small sample sizes. Therefore, we feel that there is a great need for a randomized controlled trial with an appropriate design and sample size to confirm these findings.

The aim of this study is to investigate if cCXL is non-inferior to sCXL (10 mW/cm2) in terms of flattening of the corneal surface and halting the disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Progressive keratoconus based on an increase of maximum keratometry (Kmax) of 1 diopter (D) over a time period of 12 months

Exclusion Criteria:

* Corneal scarring
* Corneal disease other than keratoconus
* History of corneal surgery (e.g. refractive surgery, corneal transplantation, intracorneal ring segments)
* Patient unwilling or unable to give informed consent, unwilling to accept randomization or inability to complete follow-up (e.g. hospital visits) or comply with study procedures
* Insufficient corneal thickness including epithelium < 375 µm
* Pregnancy
* Among patients in whom both eyes are eligible only the first eye which is undergoing corneal cross-linking is enrolled in the study
* Participation in another clinical study

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 124 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-05 (Actual)

PRIMARY OUTCOMES:
Change in maximum keratometry (Kmax) | 12 months postoperatively
  Kmax is measured with Scheimpflug photography (Pentacam® HR, OCULUS Optikgeraete GmbH, Wetzlar, Germany)

SECONDARY OUTCOMES:
Visual acuity | at baseline, 4 weeks, 3 months, 6 months and 12 months postoperatively
  Measured with ETDRS
Refraction | at baseline and 12 months postoperatively
  Change in spherical equivalent
Depth and size of demarcation line | at 4 weeks and 12 months postoperatively
  Measured with AS OCT
Pachymetry | at baseline, 4 weeks, 3 months, 6 months and 12 months postoperatively
  Measured with the Pentacam HR
Zonal Kmax | at baseline, 4 weeks, 3 months, 6 months and 12 months postoperatively
  The analysis of a 3.0 mm zone centered on Kmax measured with the Pentacam HR
DUCK score | at baseline, 4 weeks, 3 months, 6 months and 12 months postoperatively
  Dutch Crosslinking for Keratconus Score is based on changes in 5 clinical parameters that are routinely assessed: age, visual acuity, refraction error, keratometry, and subjective patient experience. Each items is scored from 0 to 2 and cutoffs are determined by clinical experience.
ABCD grading system | at baseline, 4 weeks, 3 months, 6 months and 12 months postoperatively
  Anterior radius of curvature (A), Posterior radius of curvature (B), Corneal pachymetry at thinnest point (C), Distance best corrected vision (D), and a modifier (-) for no scarring, (+) for scarring that does not obscure iris details and (++) for scarring that obscures iris details
Success/failure rate | at 12 months postoperatively
  Failure is defined as progression of the disease after CXL. Progression is defined as an increase in Kmax >1D over 12 months, an increase in K1 and/or K2 >1D over 12 months and thinning and/or an increase in the rate of corneal thickness change from the periphery to the thinnest point >10% over 12 months
Mean endothelial cell loss | at 6 and 12 months postoperatively
  Measured using specular microscopy photography
Rate of reepithelialisation | 4 days postoperatively
  evaluated with fluorescein and blue light, a slit lamp image is taking to perform quantitative morphometric surface analysis
Patient Reported Outcomes Measures (PROMs) | at baseline, 3 months, 6 months and 12 months postoperatively
  Health-related quality of life as measured by HUI3 (Health Utility Index Mark 3) questionnaire
Patient Reported Outcomes Measures (PROM) | at baseline, 3 months, 6 months and 12 months postoperatively
  Patient satisfaction and vision-specific quality of life as measured by National Eye Institute Visual Function Questionnaire (NEI VFQ-25)
Patient Reported Outcomes Measures (PROM) | at baseline, 3 months, 6 months and 12 months postoperatively
  Patient satisfaction and vision-specific quality of life as measured by Keratoconus Outcome Research Questionnaire (KORQ)
Pain after crosslinking | 4 days postoperatively
  measured with the short form of the McGill Pain Questionnaire (SF-MPQ)
Quality Adjusted Life Years (QALYs) | baseline until 12 months postoperatively
  Calculated based on generic health-related quality of life, using the EQ-5D-5L questionnaire
Quality Adjusted Life Years (QALYs) | baseline until 12 months postoperatively
  Calculated based on generic health-related quality of life, using the HUI-3 questionnaire
Costs per patient | baseline until 12 months postoperatively
  Cost per patient, including valuation of resource use by using the Dutch guidelines for cost-analyses or cost prices provided by the medical center.
Incremental cost-effectiveness ratios (ICERs): QALY | baseline until 12 months postoperatively
  Evaluation of cost-effectiveness by using calculated costs per quality-adjusted life years (QALYs)
Incremental cost-effectiveness ratios (ICERs): NEI VFQ-25 | baseline until 12 months postoperatively
  Calculated costs per clinically improved patient on the NEI VFQ-25 questionnaire
Incremental cost-effectiveness ratios (ICERs): Kmax | baseline until 12 months postoperatively
  incremental healthcare costs per patient with a reduction in Kmax of ≥ 1D after crosslinking
Incremental cost-effectiveness ratios (ICERs): visual acuity | baseline until 12 months postoperatively
  incremental healthcare costs per patient with clinical improvement in (un-) corrected distance visual acuity
Budget impact | baseline until 12 months postoperatively
  Reported as a difference in costs. Different scenario's will be compared to investigate the impact of various levels of implementation (e.g. 25%, 50%, 75% of eligible patients)

CONTACTS AND LOCATIONS:
Overall Officials: R.M.M.A. Nuijts, MD, PhD, Principal Investigator — Department of Ophthalmology, Maastricht University Medical Center (MUMC+)
Locations (3):
- Netherlands (3):
  - Maastricht University Medical Center (MUMC+), Maastricht, Limburg
  - University Medical Center Groningen, Groningen
  - University Medical Center Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Vandevenne MMS, Berendschot TTJM, Winkens B, van den Biggelaar FJHM, Visser N, Dickman MM, Wisse RPL, Wijdh RHJ, Roy AS, Shetty R, Nuijts RMMA. Efficacy of customized corneal crosslinking versus standard corneal crosslinking in patients with progressive keratoconus (C-CROSS study): study protocol for a randomized controlled trial. BMC Ophthalmol. 2023 May 19;23(1):224. doi: 10.1186/s12886-023-02976-4. PMID 37208674